CLINICAL TRIAL: NCT05136209
Title: Comparison of Posterior Continuous Curvilinear Capsulorhexis With or Without Anterior Vitrectomy in Congenital Cataract Surgery
Brief Title: Comparison of Posterior Continuous Curvilinear Capsulorhexis With or Without Anterior Vitrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCPMOH2021-China12
Record Dates: First submitted 2021-11-11; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Congenital Cataract
Keywords: Congenital cataract surgery; anterior vitrectomy; postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCCC procedure without A-vit (Experimental): Procedure/Surgery: PCCC procedure without A-vit ACCC + I / A + PCCC or ACCC + I / A +PCCC + IOL
  Interventions: Procedure: PCCC procedure without A-vit
- PCCC+A-Vit procedure (Active Comparator): Procedure/Surgery: PCCC+A-Vit procedure ACCC + I / A + PCCC + A-vit or ACCC + I / A +PCCC + IOL + A-vit
  Interventions: Procedure: PCCC+A-Vit procedure

INTERVENTIONS:
Procedure: PCCC procedure without A-vit — In this randomized clinical trial, patients receive cataract surgery on both eyes on the same day. For each patient, one eye is randomly assigned to undergo PCCC+A-Vit procedure, while the fellow eye is undergoing PCCC procedure without A-Vit.
  Arms: PCCC procedure without A-vit
Procedure: PCCC+A-Vit procedure — PCCC+A-Vit procedure
  Arms: PCCC+A-Vit procedure

SUMMARY:
Selecting the appropriate surgical approach for congenital cataracts presents challenging for ophthalmologists. This prospective, randomized controlled study aims to compare the prognosis of posterior continuous curvilinear capsulorhexis (PCCC) with or without anterior vitrectomy (A-Vit) in treating congenital cataracts.

DETAILED DESCRIPTION:
Due to the particularity of children's eye structure, selecting the appropriate surgical approach for congenital cataracts presents challenging for ophthalmologists. The major concerned postoperative problem is the after-cataract formation. As a result, PCCC with A-Vit is usually performed to prevent the formation of secondary cataracts. However. Debate over the indication and surgical procedure still persists since A-Vit and excessive manipulations may interfere with the development of the eye and increase the risk of postoperative inflammation, unstable intraocular pressure, macular edema, retinal detachment and so on. Thus, it is necessary to evaluate the safety and effectiveness of PCCC without A-Vit in congenital cataract surgery.

In this randomized clinical trial, children with equal degree of congenital cataract in both eyes are enrolled. Patients receive cataract surgery on both eyes on the same day. For each patient, one eye is randomly assigned to undergo PCCC+A-Vit procedure, while the fellow eye is undergoing PCCC procedure without A-Vit. PCCC+A-Vit procedure includes anterior continuous curvilinear capsulorhexis (ACCC), irrigation/aspiration (I/A), PCCC, and A-Vit. Primary intraocular lens implantation (IOL) is performed in children older than age of two. Investigators then compare the incidence of visual axis opacity, uveitis, iris/pupil abnormality and intraocular pressure between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Children with bilateral congenital cataracts without other ocular abnormalities
* Gestational age at birth >37 weeks
* No more than 18 years old
* Pupils could dilate normally pre-operation
* Have signed a consent form
* Can be followed

Exclusion Criteria:

* Intraocular pressure >21 mmHg
* History of ocular trauma and intraocular surgery

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with visual axis opacification | 5 years
  Number of participants with visual axis opacification evaluated based on the retro-illumination.
Number of participants with uveitis and iris/pupil abnormality | 5 years
  Number of participants with uveitis and iris/pupil abnormality evaluated based on the slip lamp examination.
IOP | 5 years
  Intraocular pressure measured by the Tono-pen or non-contact tonometer

SECONDARY OUTCOMES:
BCVA change | 5 years
  Change from baseline in the best corrected visual acuity (BCVA) measured by the Teller's acuity card, the Lea symbol visual acuity chart or the ETDRS chart according the patient's age.
AL change | 5 years
  Change from baseline in axial length measured by AL-Scan, IOLMaster or A-scan
CCT change | 5 years
  Change from baseline in the central corneal thickness (CCT) measured by pentacam.
CFT change | 5 years
  Change from baseline in the central foveal thickness (CFT) measured by Optical Coherence Tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Weirong Chen, MD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No